CLINICAL TRIAL: NCT06766903
Title: Effects of a Physical Exercise Program on Cardiovascular, Metabolic, Physical Fitness and Quality of Life in Cancer Survivors' Adult Women
Brief Title: Onco-Vascular Exer-Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristian Alvarez (Other)
Collaborators: Instituto Nacional de Deportes (Unknown)
Responsible Party: Sponsor-Investigator, Cristian Alvarez, Principal investigator, Universidad Nacional Andres Bello
Organization: Universidad Nacional Andres Bello (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UNAB-FCR-KINE2024A
Record Dates: First submitted 2024-12-26; First posted 2025-01-09 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Vascular Disease，Peripheral; Arterial Hypertension; Endothelial Dysfunction; Metabolic Disease
Keywords: Exercise training; Concurrent training; High-intensity interval training; Resistance training; Arterial stiffness; Pulse wave velocity; Carotid intima-media thickness; Flow mediated dilation; Cancer survivors; Cardiorrespiratory fitness; Physical fitness
MeSH Terms: conditions — Breast Neoplasms; Peripheral Vascular Diseases; Hypertension; Metabolic Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: It will be compared two different breast cancer survivors groups under exercise training condition, such as; exercise group of high chemotherapy (EG-HCT) or a control condition that will be an exercise group of low chemotherapy (EG-LCT).
Who Masked: Participant, Investigator
Masking Description: All participants will be randomly allocated to blinded to "participants" and "investigators" to an exercise group of high chemotherapy (EG-HCT) or a control condition that will be an exercise group of low chemotherapy (EG-LCT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EG-HCT (Experimental): (EG-HCT) Exercise group high chemotherapy dose: All participants of this groups will be breast cancer survivors and received no more than 7 chemotherapy sessions during cancer treatment.
  Interventions: Behavioral: Exercise training
- EG-LCT (Active Comparator): (EG-LCT) Exercise group low chemotherapy dose: All participants of this groups will be breast cancer survivors and received more than 8 chemotherapy sessions during cancer treatment.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — All subjects will participate of 8-weeks of exercise training intervention of concurrent training of high-intensity interval training (HIIT) using stationnaire bikes plus resistance training (RT) using free weight under lab conditions.
  The exercise program will be monitored by 8-weeks, adapted individually to each participants in terms of exercise intensity an volume.
  Other Names: Physical therapy intervention

SUMMARY:
In Chile, in the year 2022, the main causes of death were diseases of the circulatory system (31,606) and cancer (with 28,453 deaths). Both causes of death came from diseases such as arterial hypertension, diabetes, and obesity, all highly associated to sedentary lifestyle (i.e., spending long hours sitting), physical inactivity (i.e., not adhering to international recommendations of physical activity per week of 150 to 300 min of low to moderate intensity physical activity, or 75 to 150 min of vigorous physical activity per week) and others risk factors (i.e., healthy eating, and inflammation processes such as cancer). Worryingly, in the Bío-Bío, Chile region, women's deaths from cancer reported 1,380 deaths, one of the highest disease mortality in this country. On the other hand, exercise training (i.e., defined as a particular type of physical activity guided by a professional and regulated overtime) has demonstrated evidence to the prevention and treatment of cancer, as well as in diabetes and arterial hypertension (co-morbidities). This benefits of exercise training has been raised by the American College of Sports Medicine (ACSM), emphasizing the evidence in favor of the exercise training (i.e., particularly aerobic/moderate-intensity continuous and resistance-type exercise) from the strongest (anxiety, depression, fatigue, quality of life, lymphedema, physical function) to the least amount of evidence (cardio-vascular, pain, etc) benefits on cancer survivors. However, there is scarcity of knowledge about the effects of other exercise modalities such as concurrent training on cardiovascular, metabolic and physical fitness of adul woman breast cancer survivors.

DETAILED DESCRIPTION:
Despite the "solid" evidence in favor of the effects of exercise training in cancer survivors (CS) to improve variables such as anxiety, depressive symptoms, fatigue, quality of life, lymphedema, and physical function, unfortunately they are still unknown and there is minimal evidence about the effects of exercise training on cardio-vascular and metabolic variables in cancer survivors' persons. The phenomenon of the exercise training in CS persons is of relevance, because as it is pointed out, cancer is the second cause of death in Chile, and in particular breast cancer is the first cause among all types of cancer, and where exercise training has a relevant value as a treatment and post-treatment. Thus, it is required to fill the scientific gap in terms of the need to increase the evidence of exercise training in cardio-vascular physiologyof CS population, such as parameters related to blood pressure, and endothelial dysfunction such as carotid intima-media thickness (cIMT), dilation-mediated flow (FMD) and pulse wave velocity (PWV), as well as metabolic factors related to the resting metabolism and metablism during exercise such as the oxidative and glycolytic capacity, which determine the oxidation of fat and glucose during resting and exercise. There is consolidated or "solid" evidence, about the effects of physical exercise, according to the American College of Sports Medicine (ACSM) exercise recommendations guide for CS.

Different types of exercise training modalities have been reported in breast CS individuals during and following the completion of their treatment (Radiotherapy, Chemotherapy, Hormonal therapy), where the benefits of aerobic nature exercise training predominantly (i.e., exercises that promote an increase in aerobic enzymatic activity, mitochondrial biogenesis and in general oxidative metabolism [that promote the elaboration of ATP via fatty acids]) in combination with muscle strength as resistance training with the use of external overloads (i.e., controlled exercises with a certain level of muscle load based on prior assessment of maximal strength, usually measured by means of 1-repetition maximal test on different muscle groups), which are exercises that promote an increase in protein synthesis, muscle mass formation, and therefore both types of exercise training (Moderate-intensity continuous [MICT] + resistance training [RT]) are usually referred to in the literature as combined exercise or concurrent exercise (MICT+RT). Among the main effects or benefits of exercise training in breast CS individuals, particularly in terms of reducing anxiety, depressive symptoms, fatigue, quality of life, lymphedema, and physical function. It has also been reported that there is only "moderate" evidence on the effects of exercise in CS at the level of bone health, and sleep, but worryingly, there is insufficient evidence in favor of physical exercise at the level of vascular function, falls, cognitive function, and pain, among other health parameters (sexual function, nausea, peripheral neuropathies). The potential results of the project will ultimately translate into greater technical, scientific and management knowledge to be able to analyze the increase in the offer of physical exercise programs or workshops for breast CS persons in Chile. The latter should translate into an improvement not only in the physical condition and health of CS people, but also in a lower risk of relapsing into cancer, mental illnesses (depression) and, of course, a reduction in mortality. From here, high-intensity interval training, a particular exercise modality of brief intense exercise intervals have been poorly studied in breast CS. Similarly, RT using lower exercise intensities (i.e., one repetition maximum test [1RM] load of ≤60% of 1 RM) have been also little tested for cardio-vascular (i.e., PWV, FMD, and cIMT) and metabolic health in breast CS women. Preliminary evidence show that concurrent exercise training decrease blood pressure, and that high-intensity interval training (HIIT) also decrease arterial stiffness in adult women. Eight-weeks of HIIT was superior to MICT for increasing FMD in HIIT vs MICT (Δ+8.9 vs. 5.1%). Twelve-weeks of HIIT (four sets [4 min] intervals at 80-90% HRmax with resting periods of 60-70% HRmax cycling) reduced minimally PWV (-0.1 m·s-1) in hypertensive older adults. One-year of HIIT (60 s interval, 60 s of resting at 90% of the reserve oxygen consumption) decreased both systolic [SBP] (Δ-6.5)/diastolic [DBP] blood pressure (Δ-4.2 mmHg), and decreased cIMTav (Δ-0.95 mm). Thus, concurrent training of both HIIT plus RT in lower 1RM intensities could promote potential benefits for both cardiovascular health and metabolic and physical condition parameters of breast CS women, however, there is scarcity of studies about this exercise modalities in patients who are CS and that have been exposure to higher and lower chemotherapy doses.

RESEARCH PROBLEM: Despite the "solid" evidence in favor of the effects of exercise training in breast CS to improve variables such as anxiety, depressive symptoms, fatigue, quality of life, lymphedema and physical function, however, unfortunately, the effects of exercise training on cardio-vascular and metabolic variables, there is still unknown the effects of concurrent exercise training including HIIT plus RT in lower 1RM doses in CS women at level of their cardio-vascular and metabolic health. This is due to the fact that year after year there is an increase in the number of early diagnoses, as well as an increase in the number of CS with a successful completion of their breast cancer treatment (Radiotherapy, Chemotherapy, Hormonal Therapy), which also leads as an effect to an inherent increase in the number of CS persons, requiring the insertion of this population back into active life. Another effect of the scientific rationale lies in the scarce offer of physical activity and/or exercise training programs for this population of women between 40 and 70 years of age, which would be significantly overcome with the application of the present intervention project that would report cardiovascular, metabolic, physical condition, quality of life and eating patterns variables.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosed
* With/without chemotherapy treatment
* Normal weight body mass index [BMI] 18.6 to 24.9 or overweight/obesity condition by BMI 25.0 to 39.9 kg/m2
* Age 30 to 75 years
* With/without other associated co-morbidities (diagnosed of elevated fasting glucose, prediabetes or diabetes, hypertension or prehypertension, or metabolic syndrome, fatty liver or hypercholesterolemia or screened by our research team).
* With/without hormonal therapy
* With/without other pharmacotherapy for specific muscle-groups such as morphine patches, morphine droplets or other pharmacological therapy for SOS pain treatment

Exclusion Criteria:

* History of abnormal ECG
* Diagnosis of other cardio-vascular condition/history other than hypertension, vasculopathy
* History of uncontrolled stage 3 of hypertension or hypertensive crisis
* Diabetes complications such as varicose ulcers, nephropathies
* Skeletal muscle abnormalities (e.g., knee, or hip arthrosis, muscle pain)
* Using weight loss treatment/pharmacotherapy or being active in exercise training programs (or within the past three months)
* Use other pharmacotherapy that can influence body weight loss,
* Respiratory disease type (chronic obstructive disease)
* Kidney disease
* Pregnancy
* Smoking behaviour or dependence on other substances.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation in (cm) | Baseline, 8 weeks after exercise training intervention
  Change in flow-mediated dilation in the brachial artery registered by a linear transducer using images from a Doppler ultrasound
Pulse wave velocity in (m/s) | Baseline, 8 weeks after exercise training intervention
  Change in pulse wave velocity in the brachial artery registered by an oscillometric cuff in the brachial artery
Carotid intima media thickness average in (cm) | Baseline, 8 weeks after exercise training intervention
  Change in Carotid intima media thickness in the common carotid artery registered by a linear transducer using images from a Doppler ultrasound
Carotid intima media thickness maximum in (cm) | Baseline, 8 weeks after exercise training intervention
  Change in Carotid intima media thickness maximum in the common carotid artery registered by a linear transducer using images from a Doppler ultrasound

SECONDARY OUTCOMES:
Body mass in (kg) | Baseline, 8 weeks after exercise training intervention
  Change in body mass registered by a digital scale in kilograms
Body mass index in (kg/m2) | Baseline, 8 weeks after exercise training intervention
  Change in body mass index registered by from the calculation of the weight plus the height dividev by the suare of the height
Body fat in (%) | Baseline, 8 weeks after exercise training intervention
  Change in body fat percentage registered by from a digital bio-impedanciometer equipment
Skeletal muscle mass in (%) | Baseline, 8 weeks after exercise training intervention
  Change in skeletal muscle mass in percentage registered by from a digital bio-impedanciometer equipment
Resting metbolic rate in (kcal) | Baseline, 8 weeks after exercise training intervention
  Change in resting metabolic rate obtained in kcalories from a digital bio-impedanciometer equipment
Waist circumference in (cm) | Baseline, 8 weeks after exercise training intervention
  Change in waist circumference obtained from a measuring tape in centimeters
Systolic blood pressure in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in systolic blood pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position
Diastolic blood pressure in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in diastolic blood pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position
Mean arterial pressure in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in mean arterial pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position, particularly from the data systolic and diastolic blood pressure obtained from this equipment
Pulse pressure in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in pulse pressure obtained from a digital cuff sphingomanometer in mmHg from the brachial artery in seated position, particularly from the data systolic and diastolic blood pressure obtained from this equipment
Heart rate at rest in (beats/min) | Baseline, 8 weeks after exercise training intervention
  Change in heart rate at rest obtained from a digital watch cardiometer in beats/min
Systolic blood pressure of the ankle in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in systolic blood pressure obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Diastolic blood pressure of the ankle in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in systolic blood pressure obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Partial oxygen saturation in (%) | Baseline, 8 weeks after exercise training intervention
  Change in Partial oxygen saturation in (%) obtained from a digital saturometer from the index finger in seated position
Total chlesterol in (mg/dL) | Baseline, 8 weeks after exercise training intervention
  Change in total cholesterol in (mg/dL) obtained from a capillary droplet sample from the index finger from a digital portatile equipment
Fasting glucose in (mg/dL) | Baseline, 8 weeks after exercise training intervention
  Change in fasting glucose in (mg/dL) obtained from a capillary droplet sample from the index finger from a digital portatile equipment
Triglycerides in (mg/dL) | Baseline, 8 weeks after exercise training intervention
  Change in triglycerides in (mg/dL) obtained from a capillary droplet sample from the index finger from a digital portatile equipment
Lactate | Baseline, 8 weeks after exercise training intervention
  Change in Lactate in (mmol/L) obtained from a capillary droplet sample from the index finger from a digital portatile equipment
Augmentation index in (%) | Baseline, 8 weeks after exercise training intervention
  Change in Augmentation index in (%) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Ankle-Brachial Index in (%) | Baseline, 8 weeks after exercise training intervention
  Change in Ankle-Brachial Index in (%) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Aortic Systolic blood pressure in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in Aortic Systolic blood pressure in (mmHg) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Aortic pulse pressure in (mmHg) | Baseline, 8 weeks after exercise training intervention
  Change in Aortic pulse pressure in (mmHg) obtained from a digital cuff sphingomanometer in mmHg by the Arteriograpgh equipment from the brachial artery in supine position.
Aortic augmentation index in (%) | Baseline, 8 weeks after exercise training intervention
  Change in Aortic augmentation index in (%) obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Ejection duration in (m/s) | Baseline, 8 weeks after exercise training intervention
  Change in Ejection duration in (m/s) obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Diastolic reflection area | Baseline, 8 weeks after exercise training intervention
  Change in Diastolic reflection area obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Systolic area index | Baseline, 8 weeks after exercise training intervention
  Change in Diastolic area index obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Diastolic area index | Baseline, 8 weeks after exercise training intervention
  Change in Diastolic area index obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Return time of the aortic pulse wave | Baseline, 8 weeks after exercise training intervention
  Change in Return time of the aortic pulse wave measured in the brachial artery obtained from a digital cuff sphingomanometer in % by the Arteriograpgh equipment from the brachial artery in supine position.
Arterial age | Baseline, 8 weeks after exercise training intervention
  Change in arterial age estimated from a digital cuff Arteriograph equipment measured from the brachial artery
Heart rate during exercise in (beats/min) | Baseline, 8 weeks after exercise training intervention
  Heart rate measured using a cardiometer watch equipment at different power output intensities using an cycle ergometer equipment
Peak oxigen consumption (VO2peak) | Baseline, 8 weeks after exercise training intervention
  Change in VO2peak estimated from an equipment of indirect calorimetry and gas calibration of O2/VCO2, measured from breathing by breathing on a stationnaire bike ergometer
Fat oxidation (FATox) | Baseline, 8 weeks after exercise training intervention
  Change in FATox estimated from an equipment of indirect calorimetry and gas calibration of O2/VCO2, measured from breathing by breathing during 10 minutes on a stretcher
Carbohydrate oxidation (CHOox) | Baseline, 8 weeks after exercise training intervention
  Change in CHOox estimated from an equipment of indirect calorimetry and gas calibration of O2/VCO2, measured from breathing by breathing during 10 minutes on a stretcher
Maximum strength of leg extension (1RMleg) | Baseline, 8 weeks after exercise training intervention
  Change in the 1RMleg strength estimated from a leg-extension exercise machine using kilograms
Maximum strength of biceps curl (1RMbiceps) | Baseline, 8 weeks after exercise training intervention
  Change in the 1RMbiceps strength estimated using free weight in kilograms, bilateral and in stand position
Maximum strength of shoulder press (1RMsp) | Baseline, 8 weeks after exercise training intervention
  Change in the 1RMsp strength estimated using free weight in kilograms, bilateral and in stand position
Maximum strength of back exercise (1RMb) | Baseline, 8 weeks after exercise training intervention
  Change in the 1RMb strength estimated using free weight in kilograms, bilateral and in stand position

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Araneda, PhD, Study Chair — Universidad Andres Bello
Locations (1):
- ICER-Lab, Talcahuano, Chile

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT06766903/Prot_SAP_000.pdf
  • Informed Consent Form (2024-12-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT06766903/ICF_002.pdf